CLINICAL TRIAL: NCT03308318
Title: A New Discovery on the Temporal Fascial Layers: Does the Deep Layer of the Deep Temporalis Fascia Really Exist?
Brief Title: Does the Deep Layer of the Deep Temporalis Fascia Really Exist?
Status: Completed | Type: Observational
Sponsor: West China College of Stomatology (Other)
Responsible Party: Principal Investigator, Hui Li, Principal Investigator, West China College of Stomatology
Other Study IDs: hui_owe
Record Dates: First submitted 2017-10-05; First posted 2017-10-12 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Anatomy; Temporal Region Trauma
Keywords: Deep temporal fascia; Deep layer of the deep temporal fascia; Superficial layer of the deep temporal fascia; Temporal fascial layers; Temporal anatomy
MeSH Terms: conditions — Craniocerebral Trauma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the supratemporalis approach: patients operated upon with zygomaticofacial or craniofacial fractures using the supratemporalis approach
  Interventions: Procedure: The supratemporalis approach

INTERVENTIONS:
Procedure: The supratemporalis approach — The incision differs according to specific fracture sites. It can be a hockey stick-shaped incision, hemicoronal incision, and full coronal incision. The first layer of dissection was just under the superficial temporalis fascia.Then, approximately at the level of 3-5cm above the zygomatic arch, our modified incision was carried through the deep temporalis fascia.Next, the superficial fat pad was encountered and retracted anteriorly, which was in close contact of the temporal muscle. Finally, a flap that included skin, subcutaneous tissue, the superficial temporal fascia, the areolar fat tissue, the deep temporalis fascia and the superficial temporal fat was reflected as a whole anteriorly, fully exposing the temporal muscle and zygomatic arch.

SUMMARY:
It has been widely accepted that a split of the deep temporal fascia occurs approximately 2 to 3 cm above the zygomatic arch, named the superficial and deep layers. The deep layer of the deep temporal fascia lies between superficial temporal fat pad and the temporal muscle. However, during the investigators' previous surgeries, the investigators did not find the deep layer of the deep temporal fascia between superficial temporal fat pad and the temporal muscle. This study was conducted to clarify the presence or absence of the deep layer of the deep temporal fascia. And the investigators' clinical study has confirmed the absence of the deep layer of the deep temporal fascia between superficial temporal fat pad and the temporal muscle.

DETAILED DESCRIPTION:
The anatomic layers of soft tissues of the temporal region, with regard to the deep temporalis fascia, was investigated in 169 cases operated upon with zygomaticofacial or craniofacial fractures using the supratemporalis approach from June 2013 to June 2017. Among 167 surgeries, this so-called "deep layer of the deep temporalis fascia" was not observed. In fact, the superficial temporal fat pad is closely attached to temporal muscle above the zygomatic arch.

ELIGIBILITY:
Inclusion Criteria:

Clinical and imaging diagnosis of zygomaticofacial or craniofacial fractures A need to operate using the supratemporalis approach No previously surgical treatment

Exclusion Criteria:

unobvious displaced fracture disagree with the surgical treatment previous unsuccessful surgery at the temporal region

Ages: 10 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients diagnosed with zygomaticofacial fractures or craniofacial fractures and received surgical treatment from the Dr. Lei Liu
Sampling Method: Probability Sample
Enrollment: 167 (Actual)
Dates: Start 2013-06-17 (Actual); Primary Completion 2017-06-13 (Actual); Study Completion 2017-06-13 (Actual)

PRIMARY OUTCOMES:
deep layer of the deep temporal fascia | during surgery
  the investigators did not find the deep layer of the deep temporal fascia between superficial temporal fat pad and the temporal muscle

CONTACTS AND LOCATIONS:
Overall Officials: Lei Liu, DMD, Study Director — Department of Oral & Maxillofacial Surgery, West China Hospital of Stomatology, Sichuan University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krayenbuhl N, Isolan GR, Hafez A, Yasargil MG. The relationship of the fronto-temporal branches of the facial nerve to the fascias of the temporal region: a literature review applied to practical anatomical dissection. Neurosurg Rev. 2007 Jan;30(1):8-15; discussion 15. doi: 10.1007/s10143-006-0053-5. Epub 2006 Nov 10. PMID 17096156
- [Background] O'Brien JX, Ashton MW. Relationship of the temporofrontal rami of the facial nerve to the fascial layers of the temporal region. Ann Plast Surg. 2012 Jun;68(6):547-8. doi: 10.1097/SAP.0b013e318221b563. PMID 22643100
- [Background] Ammirati M, Spallone A, Ma J, Cheatham M, Becker D. An anatomicosurgical study of the temporal branch of the facial nerve. Neurosurgery. 1993 Dec;33(6):1038-43; discussion 1044. doi: 10.1227/00006123-199312000-00012. PMID 8133989
- [Background] Agarwal CA, Mendenhall SD 3rd, Foreman KB, Owsley JQ. The course of the frontal branch of the facial nerve in relation to fascial planes: an anatomic study. Plast Reconstr Surg. 2010 Feb;125(2):532-537. doi: 10.1097/PRS.0b013e3181c82e9d. PMID 20124839
- [Background] Tellioglu AT, Tekdemir I, Erdemli EA, Tuccar E, Ulusoy G. Temporoparietal fascia: an anatomic and histologic reinvestigation with new potential clinical applications. Plast Reconstr Surg. 2000 Jan;105(1):40-5. doi: 10.1097/00006534-200001000-00007. PMID 10626968
- [Background] Coscarella E, Vishteh AG, Spetzler RF, Seoane E, Zabramski JM. Subfascial and submuscular methods of temporal muscle dissection and their relationship to the frontal branch of the facial nerve. Technical note. J Neurosurg. 2000 May;92(5):877-80. doi: 10.3171/jns.2000.92.5.0877. PMID 10794306
- [Background] Wormald PJ, Alun-Jones T. Anatomy of the temporalis fascia. J Laryngol Otol. 1991 Jul;105(7):522-4. doi: 10.1017/s0022215100116500. PMID 1875131
- [Background] Stuzin JM, Wagstrom L, Kawamoto HK, Wolfe SA. Anatomy of the frontal branch of the facial nerve: the significance of the temporal fat pad. Plast Reconstr Surg. 1989 Feb;83(2):265-71. doi: 10.1097/00006534-198902000-00011. PMID 2911626
- [Background] Abul-Hassan HS, von Drasek Ascher G, Acland RD. Surgical anatomy and blood supply of the fascial layers of the temporal region. Plast Reconstr Surg. 1986 Jan;77(1):17-28. PMID 3941846
- [Background] Tolhurst DE, Carstens MH, Greco RJ, Hurwitz DJ. The surgical anatomy of the scalp. Plast Reconstr Surg. 1991 Apr;87(4):603-12; discussion 613-4. PMID 2008459
- [Background] Ramirez OM. Endoscopic techniques in facial rejuvenation: an overview. Part I. Aesthetic Plast Surg. 1994 Spring;18(2):141-7. doi: 10.1007/BF00454473. PMID 8017216
- [Background] Stuzin JM, Baker TJ, Gordon HL. The relationship of the superficial and deep facial fascias: relevance to rhytidectomy and aging. Plast Reconstr Surg. 1992 Mar;89(3):441-9; discussion 450-1. PMID 1741467
- [Background] Accioli de Vasconcellos JJ, Britto JA, Henin D, Vacher C. The fascial planes of the temple and face: an en-bloc anatomical study and a plea for consistency. Br J Plast Surg. 2003 Oct;56(7):623-9. doi: 10.1016/s0007-1226(03)00310-2. PMID 12969659
- [Background] Campiglio GL, Candiani P. Anatomical study on the temporal fascial layers and their relationships with the facial nerve. Aesthetic Plast Surg. 1997 Mar-Apr;21(2):69-74. doi: 10.1007/s002669900086. PMID 9143418
- [Background] Rowe NL. Surgery of the temporomandibular joint. Proc R Soc Med. 1972 Apr;65(4):383-8. doi: 10.1177/003591577206500438. No abstract available. PMID 5024527
- [Background] Al-Kayat A, Bramley P. A modified pre-auricular approach to the temporomandibular joint and malar arch. Br J Oral Surg. 1979 Nov;17(2):91-103. doi: 10.1016/s0007-117x(79)80036-0. PMID 298842
- [Background] Politi M, Toro C, Cian R, Costa F, Robiony M. The deep subfascial approach to the temporomandibular joint. J Oral Maxillofac Surg. 2004 Sep;62(9):1097-102. doi: 10.1016/j.joms.2003.10.013. PMID 15346360
- [Background] Candirli C, Celik S. Efficacy of deep subfascial approach to the temporomandibular joint. J Craniofac Surg. 2012 Mar;23(2):e126-9. doi: 10.1097/SCS.0b013e31824cdb5c. PMID 22446445
- [Background] Nellestam P, Eriksson L. Preauricular approach to the temporomandibular joint: a postoperative follow-up on nerve function, hemorrhage and esthetics. Swed Dent J. 1997;21(1-2):19-24. PMID 9178446
- [Background] Gosain AK, Sewall SR, Yousif NJ. The temporal branch of the facial nerve: how reliably can we predict its path? Plast Reconstr Surg. 1997 Apr;99(5):1224-33; discussion 1234-6. doi: 10.1097/00006534-199704001-00003. PMID 9105349
- [Background] Hochberg J, Kaufman H, Ardenghy M. Saving the frontal branch during a low fronto-orbital approach. Aesthetic Plast Surg. 1995 Mar-Apr;19(2):161-3. doi: 10.1007/BF00450252. PMID 7598027
- [Background] Kenkere D, Srinath KS, Reddy M. Deep subfascial approach to the temporal area. J Oral Maxillofac Surg. 2013 Feb;71(2):382-8. doi: 10.1016/j.joms.2012.04.019. Epub 2012 Jun 16. PMID 22705217
- [Background] Li H, Zhang G, Cui J, Liu W, Dilxat D, Liu L. A Modified Preauricular Approach for Treating Intracapsular Condylar Fractures to Prevent Facial Nerve Injury: The Supratemporalis Approach. J Oral Maxillofac Surg. 2016 May;74(5):1013-22. doi: 10.1016/j.joms.2015.12.013. Epub 2016 Jan 7. PMID 26844401
- [Background] Babakurban ST, Cakmak O, Kendir S, Elhan A, Quatela VC. Temporal branch of the facial nerve and its relationship to fascial layers. Arch Facial Plast Surg. 2010 Jan-Feb;12(1):16-23. doi: 10.1001/archfacial.2009.96. PMID 20083736
- [Background] Kim S, Matic DB. The anatomy of temporal hollowing: the superficial temporal fat pad. J Craniofac Surg. 2005 Sep;16(5):760-3. doi: 10.1097/01.scs.0000180010.83480.10. PMID 16192853
- [Background] Tremolada C, Candiani P, Signorini M, Vigano M, Donati L. The surgical anatomy of the subcutaneous fascial system of the scalp. Ann Plast Surg. 1994 Jan;32(1):8-14. doi: 10.1097/00000637-199401000-00002. PMID 8141539
- [Background] Ramirez OM, Maillard GF, Musolas A. The extended subperiosteal face lift: a definitive soft-tissue remodeling for facial rejuvenation. Plast Reconstr Surg. 1991 Aug;88(2):227-36; discussion 237-8. PMID 1852815
- [Background] Kadri PA, Al-Mefty O. The anatomical basis for surgical preservation of temporal muscle. J Neurosurg. 2004 Mar;100(3):517-22. doi: 10.3171/jns.2004.100.3.0517. PMID 15035289
- [Background] Davidge KM, van Furth WR, Agur A, Cusimano M. Naming the soft tissue layers of the temporoparietal region: unifying anatomic terminology across surgical disciplines. Neurosurgery. 2010 Sep;67(3 Suppl Operative):ons120-9; discussion ons129-30. doi: 10.1227/01.NEU.0000383132.34056.61. PMID 20679939